CLINICAL TRIAL: NCT01616121
Title: Preemptive Lung Impedance-Guided Therapy in Evolving Acute Heart Failure in Acute Myocardial Infarction Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0037-12-HYMC
Record Dates: First submitted 2012-05-31; First posted 2012-06-11 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: In this study the interventional group was treated preemptively according to the lung-impedance protocol and the control group was treated only according to clinical assessment.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Treatment Heart Failure (Active Comparator): Conventional Treatment
  Interventions: Other: Usual treatment of patients with developing acute heart failure
- Lung Impedance-Guided Therapy (Experimental): Lung Impedance-Guided Therapy
  Interventions: Device: Lung Impedance-Guided Therapy

INTERVENTIONS:
Other: Usual treatment of patients with developing acute heart failure
  Arms: Conventional Treatment Heart Failure
Device: Lung Impedance-Guided Therapy — Non-invasive lung impedance monitor (RSMM Company, Tel Aviv, Israel)
  Arms: Lung Impedance-Guided Therapy

SUMMARY:
It is well-known that 20-25% of patients hospitalized for acute myocardial infarction will develop acute heart failure during their hospitalization. Currently, the investigators have no reliable parameter for prediction of evolving acute heart failure in such a group of patients. As a result, the investigators have no way of preventing acute heart failure. Treatment of these patients only begins after appearance of clinical signs of acute heart failure. Lung impedance monitoring may be a good non-invasive parameter for prediction of evolving acute heart failure. This study will attempt to address whether preemptive lung impedance-guided therapy may prevent the development of overt acute heart failure and improve their clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the ICCU for acute myocardial infarction and developing acute heart failure

Exclusion Criteria:

* Patients with acute myocardial infarction with clinical and radiological signs of acute heart failure at admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2002-06-01 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2014-07-01 (Actual)

PRIMARY OUTCOMES:
Prevention of acute heart failure development in acute MI patients | Three years

SECONDARY OUTCOMES:
Improvement of clinical outcome in patients with lung impedance-guided treatments | Three years

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel